CLINICAL TRIAL: NCT01961609
Title: Secukinumab In Patients With Moderate to Severe Active, Chronic Plaque Psoriasis Who Have Failed on TNFα antaGoNists: A Clinical Trial EvalUating Treatment REsults
Brief Title: Secukinumab in Tumor Necrosis Factor (TNF) - Inadequate Response (IR) Psoriasis Participants.
Acronym: SIGNATURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457AGB01
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-12

CONDITIONS: Psoriasis
Keywords: Chronic plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab (AIN457) 300 mg (Experimental): Participants self-administered 300 mg secukinumab loading dose subcutaneously at Day 0 (initiation of study drug) and at weeks 1, 2, 3 & 4, and then every 4 weeks. Following the Primary Endpoint at 16 weeks, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 32 weeks. Participants not meeting this NICE criterion returned to routine treatment under the care of their usual Clinical Team. Following assessment at week 48, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 24 weeks. Participants not meeting this NICE criterion returned to routine treatment under the care of their usual Clinical Team.
  Interventions: Biological: Secukinumab (AIN457)
- Secukinumab (AIN457) 150 mg (Experimental): Participants self-administered secukinumab 150 mg loading dose subcutaneously at Day 0 (initiation of study drug), weeks 1, 2, 3 & 4 and then every 4 weeks. Following the Primary Endpoint at 16 weeks, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 32 weeks at the 150mg dose. Participants not achieving the NICE criteria at the Primary Endpoint were up titrated to 300mg. Following assessment at week 48, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 24 weeks at the 150mg dose. Participants not achieving the NICE criteria at 48 weeks on the 150mg dose were up titrated to 300mg.
  Interventions: Biological: Secukinumab (AIN457)

INTERVENTIONS:
Biological: Secukinumab (AIN457) — Secukinumab was supplied in 150mg pre-filled syringes.

SUMMARY:
This study was designed to prove and quantify the hypothesis that secukinumab is effective, safe and well tolerated in the treatment of moderate to severe chronic plaque-type psoriasis in patients who are inadequate responders to anti-TNFα therapy in a United Kingdom (UK) and Republic of Ireland) specific population.

DETAILED DESCRIPTION:
There is no clear evidence or guidelines on appropriate treatment once a patient with moderate/severe psoriasis has failed to respond to anti-TNFα therapy, whether a single anti-TNFα therapy failure or multiple anti-TNFα therapy failures.

Numerous double-blind, double-dummy, randomised, parallel-group, active and placebo controlled studies have already been designed and run for the Phase III secukinumab clinical development program, in accordance with Health Authorities guidelines and feedback, including Food and Drug Administration (FDA) and European Medicines Agency (EMA). None of these specifically studied patients who have failed to respond to anti-TNFα therapy as defined by National Institute for Health and Care Excellence (NICE) guidelines.

Therefore, this study utilises a pragmatic, open-label, non-comparator design, which has been shown to be appropriate in similar studies looking at anti-TNFα therapy in patients failing on other therapies (Papp et al. 2012; Strober et al. 2011), to answer the question of whether secukinumab is an appropriate choice in patients who have failed to respond to anti-TNFα therapy (TNF-IR) per NICE definitions, whether a single anti-TNFα therapy failure or multiple anti-TNFα therapy failures.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed
2. Aged at least 18 years at screening
3. Chronic plaque-type psoriasis diagnosed for at least 6 months prior to screening
4. Moderate to severe disease severity:

   * PASI ≥10 and
   * DLQI >10
5. Failed to respond to systemic therapies including cyclosporine and/or methotrexate and/or PUVA (or is intolerant and/or has a contraindication to these)
6. Previously treated with at least one anti-TNFα for moderate or severe psoriasis but is a primary or secondary non-responder
7. Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Key Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis)
2. Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium)
3. Ongoing use of prohibited psoriasis treatments (e.g., topical or systemic corticosteroids (CS), UV therapy). Washout periods detailed in the protocol must be adhered to.
4. Ongoing use of other non-psoriasis prohibited treatments. Washout periods detailed in the protocol have to be adhered to. All other prior non-psoriasis concomitant treatments must be on a stable dose for at least four weeks before initiation of study drug.
5. Previous exposure to secukinumab or any other biologic drug directly targeting IL-17 or the IL-17 receptor
6. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
7. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant unless they use 2 (two) effective forms of contraception during the study and for 16 weeks after stopping treatment.
8. Men with a female partner of child bearing potential defined as all women physiologically capable of becoming pregnant unless they use 1 (one) effective form of contraception during the study and for 16 weeks after stopping treatment.
9. Active systemic infections during the last two weeks (exception: common cold) prior to initiation of study drug and any infections that reoccur on a regular basis; investigator discretion should be used regarding patients who have travelled or recently resided in areas of endemic mycoses, such as histoplasmosis, coccidioidomycosis or blastomycosis and for patients with underlying conditions that may predispose them to infection, such as advanced or poorly controlled diabetes
10. History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold test (QFT) at screening. Patients with a positive QFT test may participate in the study if further work up establishes conclusively that the patient has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment must have been initiated and maintained according to UK guidelines.
11. Known infection with HIV, hepatitis B or hepatitis C at screening or at initiation of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2016-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- Ireland (2):
  - Novartis Investigative Site, Cork
  - Novartis Investigative Site, Dublin
- United Kingdom (48):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Harlow, Essex
  - Novartis Investigative Site, London, GBR
  - Novartis Investigative Site, Canterbury, Kent
  - Novartis Investigative Site, Dafen, Llanelli
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Cliftonville, Northampton
  - Novartis Investigative Site, Nottingham, Nottinghamshire
  - Novartis Investigative Site, Aberdeen, Scotland
  - Novartis Investigative Site, Yeovil, Somerset
  - Novartis Investigative Site, Cardiff, South Glamorgan
  - Novartis Investigative Site, Staffordshire, Staffordshire
  - Novartis Investigative Site, Ipswich, Suffolk
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, Surrey, Surrey
  - Novartis Investigative Site, Rhyl, Wales
  - Novartis Investigative Site, Coventry, Warwickshire
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Airdrie
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Chester
  - Novartis Investigative Site, Durham
  - Novartis Investigative Site, Fife
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, Lancaster
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Middlesex
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Poole
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Scaroborough
  - Novartis Investigative Site, Scunthorpe
  - Novartis Investigative Site, Stoke-on-Trent
  - Novartis Investigative Site, Surrey
  - Novartis Investigative Site, Wrexham
  - Novartis Investigative Site, York

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 3 periods: initiation, maintenance 1 and maintenance 2. During the initiation period, participants received secukinumab 150 mg or 300 mg for 16 weeks.
Pre-assignment Details: For both maintenance periods 1 and 2, after 16 weeks and 48 weeks, respectively, responders at both the 150 mg and 300 mg doses continued on their initiation doses during maintenance periods 1 and 2. Non-responders at 150 mg were uptitrated to 300 mg. Non-responders at 300 mg returned to routine treatment under the care of their usual clinician.
Groups:
- Secukinumab (AIN457) 300 mg: Participants self-administered 300 mg secukinumab loading dose subcutaneously at Day 0 (initiation of study drug) and at weeks 1, 2, 3 & 4, and then every 4 weeks. Following the Primary Endpoint at 16 weeks, participants meeting the National Institute for Health and Care Excellence (NICE) criteria of adequate response were eligible to continue on study treatment for a further 32 weeks. Participants not meeting this NICE criterion returned to routine treatment under the care of their usual Clinical Team. Following assessment at week 48, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 24 weeks. Participants not meeting this NICE criterion returned to routine treatment under the care of their usual Clinical Team.
- Secukinumab (AIN457) 150 mg: Participants self-administered secukinumab 150 mg loading dose subcutaneously at Day 0 (initiation of study drug), weeks 1, 2, 3 & 4 and then every 4 weeks. Following the Primary Endpoint at 16 weeks, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 32 weeks at the 150mg dose. Participants not achieving the NICE criteria at the Primary Endpoint were up titrated to 300mg at the discretion of the treating physician. Following assessment at week 48, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 24 weeks at the 150mg dose. Participants not achieving the NICE criteria at 48 weeks on the 150mg dose were up titrated to 300mg at the discretion of the treating physician.
- Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1): Non-responders at secukinumab 150mg from the initiation period were uptitrated to secukinumab 300 mg at week 16.
- Secukinumab (AIN457) 150 mg - 300 mg (Maintenance Period 2): Non-responders at secukinumab 150 mg from maintenance 1 period were uptitrated to secukinumab 300 mg at week 48.
Period: Initiation
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1) | Secukinumab (AIN457) 150 mg - 300 mg (Maintenance Period 2)
Started | 119 | 116 | 0 | 0
Safety Set | 118 | 115 | 0 | 0
Full Analysis Set | 118 | 115 | 0 | 0
Completed | 107 | 103 | 0 | 0
Not Completed | 12 | 13 | 0 | 0
Not completed — Missing | 3 | 2 | 0 | 0
Not completed — Protocol deviation | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Administrative problems | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0
Not completed — Abnormal lab values | 0 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 5 | 0 | 0
Not completed — Randomized but not treated | 1 | 1 | 0 | 0
Period: Maintenance 1 (Weeks 17 - 48)
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1) | Secukinumab (AIN457) 150 mg - 300 mg (Maintenance Period 2)
Started | 107 | 66 | 37 | 0
Full Analysis Set | 107 | 66 | 37 | 0
Safety Set | 107 | 66 | 37 | 0
Completed | 84 | 55 | 18 | 0
Not Completed | 23 | 11 | 19 | 0
Not completed — Reason for discontinuation is missing | 1 | 0 | 3 | 0
Not completed — Protocol deviation | 3 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 13 | 4 | 10 | 0
Not completed — Adverse Event | 6 | 6 | 3 | 0
Not completed — Abnormal laboratory value | 0 | 0 | 1 | 0
Period: Maintanence 2 (Weeks 49 - 72)
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1) | Secukinumab (AIN457) 150 mg - 300 mg (Maintenance Period 2)
Started | 83 | 31 | 16 | 24
Safety Set | 83 | 31 | 16 | 24
Full Analysis Set | 83 | 31 | 16 | 24
Completed | 71 | 25 | 12 | 17
Not Completed | 12 | 6 | 4 | 7
Not completed — Reason for discontinuation is missing | 7 | 5 | 0 | 4
Not completed — Protocol deviation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Total
Number analyzed (Participants) | 119 | 116 | 235
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (11.63) | 44.6 (11.73) | 45.6 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 103
  Male | 68 | 64 | 132

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Secukinumab 300 mg Participants Achieving PASI 75 at 16 Weeks
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 75 is defined as participants achieving ≥ 75% improvement from baseline.
Time Frame: 16 weeks
Population: The full analysis set was analyzed. Missing values with respect to response variables based on PASI score have been imputed with non-response throughout regardless of the reason for missing data (e.g. premature study discontinuation, missed visit, administrative issues).
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg
Number analyzed (Participants) | 118
Percentage of participants | 65.3
Statistical Analysis 1: Comparison: Secukinumab (AIN457) 300 mg; Test type: Superiority or Other; p < 0.0001, two-sided binomial exact test; Percentage = 65.3, 99.375% CI 2-sided [52.4 to 76.7] — A Bonferroni adjustment adjusting for 8 analyses have been applied

2. Secondary Outcome: Percentage of Secukinumab 150 mg Participants Achieving PASI 75 at 16 Weeks
Description: as for outcome 1
Time Frame: 16 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 150 mg
Number analyzed (Participants) | 115
Percentage of participants | 44.3

3. Secondary Outcome: Percentage of Participants Achieving PASI 75 According to 3 Key Participant Subgroups (Primary Inadequate Response (IR), Secondary IR and IR After More Than One Anti-TNFalpha Therapies) at 16 Weeks
Description: as for outcome 1
Time Frame: 16 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Secukinumab (AIN457) 300 mg Subgroup 1; Secukinumab (AIN457) 150 mg Subgroup 1: Participants who had experienced an IR after trying the first anti-tumor necrosis factor-alpha (TNFalpha) therapy
- Secukinumab (AIN457) 300 mg Subgroup 2; Secukinumab (AIN457) 150 mg Subgroup 2: Participants who had initially experienced an adequate response after trying the first TNFalpha therapy, but then subsequently lost that response
- Secukinumab (AIN457) 300 mg Subgroup 3; Secukinumab (AIN457) 150 mg Subgroup 3: All participants who have tried and failed more than one anti-TNFalpha therapies
Arm/Group | Secukinumab (AIN457) 300 mg Subgroup 1 | Secukinumab (AIN457) 300 mg Subgroup 2 | Secukinumab (AIN457) 300 mg Subgroup 3 | Secukinumab (AIN457) 150 mg Subgroup 1 | Secukinumab (AIN457) 150 mg Subgroup 2 | Secukinumab (AIN457) 150 mg Subgroup 3
Number analyzed (Participants) | 14 | 44 | 44 | 18 | 42 | 37
Percentage of participants | 71.4 | 70.5 | 47.7 | 38.9 | 61.9 | 32.4

4. Secondary Outcome: Percentage of Participants Achieiving PASI 75 - Initiation Period
Description: as for outcome 1
Time Frame: 2 ,4, 8, 12 and 16 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg
Number analyzed (Participants) | 118 | 115
Percentage of participants
  Week 2 | 1.7 | 2.6
  Week 4 | 27.1 | 18.3
  Week 8 | 60.2 | 40.0
  Week 12 | 61.9 | 52.2
  Week 16 | 65.3 | 44.3

5. Secondary Outcome: Percentage of Participants Achieiving PASI 75 - Maintenance 1 Period
Description: as for outcome 1
Time Frame: 16, 24 and 48 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1)
Number analyzed (Participants) | 107 | 66 | 37
Percentage of participants
  Week 16 | 72.0 | 75.8 | 2.7
  Week 24 | 61.7 | 68.2 | 13.5
  Week 48 | 52.3 | 39.4 | 8.1

6. Secondary Outcome: Percentage of Participants Achieiving PASI 75 - Maintenance 2 Period
Description: as for outcome 1
Time Frame: 48 and 72 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1) | Secukinumab (AIN457) 150 mg - 300 mg (Maintenance Period 2)
Number analyzed (Participants) | 83 | 31 | 16 | 24
Percentage of participants
  Week 48 | 65.1 | 80.6 | 18.8 | 4.2
  Week 72 | 65.1 | 58.1 | 25.0 | 37.5

7. Secondary Outcome: Percentage of Participants Achieving PASI 50 and PASI 90 - Initiation Period
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 50 and PASI 90 are defined as participants achieving ≥ 50% and ≥ 90% improvement from baseline, respectively.
Time Frame: 2, 4, 8, 12, 16 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg
Number analyzed (Participants) | 118 | 115
Percentage of participants
  PASI 50, week 2 | 28.0 | 25.2
  PASI 50, week 4 | 63.6 | 57.4
  PASI 50, week 8 | 84.7 | 67.8
  PASI 50, week 12 | 82.2 | 69.6
  PASI 50, week 16 | 82.2 | 65.2
  PASI 90, week 2 | 0 | 0
  PASI 90, week 4 | 6.8 | 4.3
  PASI 90, week 8 | 25.4 | 20.0
  PASI 90, week 12 | 38.1 | 25.2
  PASI 90, week 16 | 41.5 | 20.0

8. Secondary Outcome: Percentage of Participants Achieving PASI 50 and PASI 90 - Maintenance 1 Period
Description: as for outcome 7
Time Frame: 16, 24 and 48 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1)
Number analyzed (Participants) | 107 | 66 | 37
Percentage of participants
  PASI 50, week 16 | 89.7 | 95.5 | 24.3
  PASI 50, week 24 | 80.4 | 89.4 | 54.1
  PASI 50, week 48 | 70.1 | 65.2 | 32.4
  PASI 90, week 16 | 45.8 | 34.8 | 0
  PASI 90, week 24 | 39.3 | 37.9 | 2.7
  PASI 90, week 48 | 31.8 | 18.2 | 5.4

9. Secondary Outcome: Percentage of Participants Achieving PASI 50 and PASI 90 - Maintenance 2 Period
Description: as for outcome 7
Time Frame: 48 and 72 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1) | Secukinumab (AIN457) 150 mg - 300 mg (Maintenance Period 2)
Number analyzed (Participants) | 83 | 31 | 16 | 24
Percentage of participants
  PASI 50, week 48 | 88.0 | 96.8 | 75.0 | 50.0
  PASI 50, week 72 | 74.7 | 80.6 | 37.5 | 70.8
  PASI 90, week 48 | 41.0 | 38.7 | 12.5 | 0
  PASI 90, week 72 | 38.6 | 22.6 | 18.8 | 16.7

10. Secondary Outcome: Percentage of Participants Who Have Failed on One Anti-TNFα Achieving PASI 75 (Subgroups 1 and 2 Combined) at 16 Weeks
Description: as for outcome 1
Time Frame: 16 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Secukinumab (AIN457A) 300 mg Subgroups 1 and 2 Combined); Secukinumab (AIN457) 150 mg Subgroups 1 and 2: Participants who experienced an IR after trying first anti-TNFalpha therapy and participants who had initially experienced an adequate response after trying the first anti-TNFalpha therapy but then had subsequently lost that response.
Arm/Group | Secukinumab (AIN457A) 300 mg Subgroups 1 and 2 Combined) | Secukinumab (AIN457) 150 mg Subgroups 1 and 2
Number analyzed (Participants) | 58 | 60
Percentage of participants | 70.7 | 55.0

11. Secondary Outcome: Percentage of Participants Achieving NICE Continuation Criteria (PASI 75 or PASI 50 Plus a 5 Point Improvement in DLQI) at 16 Weeks
Description: PASI 75 is defined as participants achieving ≥ 75% improvement from baseline. The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases. The measure is widely used: it has been tested across 32 different skin conditions and is available in 55 languages. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment.
Time Frame: 16 Weeks
Population: The full analysis set was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg
Number analyzed (Participants) | 118 | 115
Percentage of participants | 81.4 | 60.9

12. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI) Total Scores - Initiation Period
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases. The measure is widely used: it has been tested across 32 different skin conditions and is available in 55 languages. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment. A negative change from baseline indicates improvement.
Time Frame: Baseline, week 12, and week 16
Population: The full analysis set was considered for the analysis. Only participants who had both baseline and post baseline measurements for a given time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg
Number analyzed (Participants) | 118 | 115
score on a scale
  Week 12, initiation: number analyzed (Participants) | 111 | 108
  Week 12, initiation | -15.6 (7.49) | -13.2 (7.36)
  Week 16, initiation: number analyzed (Participants) | 109 | 103
  Week 16, initiation | -16.1 (6.80) | -12.3 (7.68)

13. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI)Total Scores - Maintenance 1 Period
Description: as for outcome 12
Time Frame: Baseline, 16, 24 and 48 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1)
Number analyzed (Participants) | 107 | 66 | 37
score on a scale
  Week 16, maintenance 1: number analyzed (Participants) | 106 | 64 | 36
  Week 16, maintenance 1 | -16.3 (6.67) | -15.9 (6.31) | -6.1 (5.86)
  Week 24, maintenance 1: number analyzed (Participants) | 102 | 64 | 35
  Week 24, maintenance 1 | -15.7 (7.25) | -14.4 (6.73) | -8.7 (6.01)
  Week 48, maintenance 1: number analyzed (Participants) | 86 | 55 | 19
  Week 48, maintenance 1 | -16.2 (8.06) | -11.5 (8.14) | -9.8 (6.76)

14. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI)Total Scores - Maintenance 2 Period
Description: as for outcome 12
Time Frame: Baseline, 48 and 72 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1) | Secukinumab (AIN457) 150 mg - 300 mg (Maintenance Period 2)
Number analyzed (Participants) | 83 | 31 | 16 | 24
score on a scale
  Week 48, maintenance 2: number analyzed (Participants) | 79 | 30 | 16 | 24
  Week 48, maintenance 2 | -17.2 (7.33) | -14.7 (6.19) | -11.5 (5.98) | -7.7 (8.80)
  Week 72, maintenance 2: number analyzed (Participants) | 74 | 26 | 12 | 21
  Week 72, maintenance 2 | -17.0 (7.27) | -13.0 (5.62) | -11.3 (4.77) | -15.0 (8.76)

15. Secondary Outcome: Mean Percent Change in EuroQOL 5-Dimension Health Status Questionnaire (EQ-5D) Health State Assessment Scores (From 0 to 100) - Initiation Period
Description: The EQ-5D is an instrument used to assess a participant's health status. The instrument includes a descriptive profile and a visual analog scale (VAS). The descriptive profile includes 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension had 3 response levels: no problems, some problems and severe problems. The VAS is a vertical scale that assesses the health status from 0 (worst possible health state) to 100 (best possible health state). This outcome measures the percent change in VAS score.
Time Frame: Baseline, 12 and 16 weeks
Population: The full analysis set was considered for the analysis. Only participants with measurements at each given time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg
Number analyzed (Participants) | 118 | 115
percent change
  Week 12, initiation: number analyzed (Participants) | 110 | 106
  Week 12, initiation | 76.25 (18.612) | 72.92 (20.004)
  Week 16, initiation: number analyzed (Participants) | 108 | 103
  Week 16, initiation | 76.30 (21.580) | 75.25 (19.100)

16. Secondary Outcome: Mean Percent Change in EuroQOL 5-Dimension Health Status Questionnaire (EQ-5D) Health State Assessment Scores (From 0 to 100) - Maintenance 1 Period
Description: as for outcome 15
Time Frame: Baseline, 16, 24 and 48 weeks
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1)
Number analyzed (Participants) | 107 | 66 | 37
percent change
  Week 16, maintenance 1: number analyzed (Participants) | 105 | 64 | 37
  Week 16, maintenance 1 | 77.33 (20.665) | 80.48 (16.099) | 67.03 (20.657)
  Week 24, maintenance 1: number analyzed (Participants) | 102 | 64 | 35
  Week 24, maintenance 1 | 79.16 (18.587) | 80.05 (16.345) | 69.14 (19.587)
  Week 48, maintenance 1: number analyzed (Participants) | 86 | 55 | 19
  Week 48, maintenance 1 | 77.73 (21.598) | 76.07 (20.413) | 70.37 (18.038)

17. Secondary Outcome: Mean Percent Change in EuroQOL 5-Dimension Health Status Questionnaire (EQ-5D) Health State Assessment Scores (From 0 to 100) - Maintenance 2 Period
Description: as for outcome 15
Time Frame: Baseline, 48 and 72 weeks
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Secukinumab (AIN457) 300 mg | Secukinumab (AIN457) 150 mg | Secukinumab (AIN457) 150 mg - 300 mg (Maintanence Period 1) | Secukinumab (AIN457) 150 mg - 300 mg (Maintenance Period 2)
Number analyzed (Participants) | 83 | 31 | 16 | 24
percent change
  Week 48, maintenance 2 (n=79,30,16,24): number analyzed (Participants) | 79 | 30 | 16 | 24
  Week 48, maintenance 2 (n=79,30,16,24) | 80.22 (19.200) | 83.87 (11.337) | 74.50 (14.855) | 67.63 (24.912)
  Week 72, maintenance 2 (n=73,26,12,21): number analyzed (Participants) | 73 | 26 | 12 | 21
  Week 72, maintenance 2 (n=73,26,12,21) | 78.24 (19.792) | 80.88 (17.635) | 77.67 (16.615) | 79.67 (18.680)

ADVERSE EVENTS:
Groups:
- Secukinumab (AIN457) 150mg: Participants self-administered secukinumab 150 mg loading dose subcutaneously at Day 0 (initiation of study drug), weeks 1, 2, 3 & 4 and then every 4 weeks. Following the Primary Endpoint at 16 weeks, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 32 weeks at the 150mg dose. Participants not achieving the NICE criteria at the Primary Endpoint were up titrated to 300mg at the discretion of the treating physician. Following assessment at week 48, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 24 weeks at the 150mg dose. Participants not achieving the NICE criteria at 48 weeks on the 150mg dose were up titrated to 300mg at the discretion of the treating physician.
- Secukinumab (AIN457) 300mg: Participants self-administered 300 mg secukinumab loading dose subcutaneously at Day 0 (initiation of study drug) and at weeks 1, 2, 3 & 4, and then every 4 weeks. Following the Primary Endpoint at 16 weeks, participants meeting the National Institute for Health and Care Excellence (NICE) criteria of adequate response were eligible to continue on study treatment for a further 32 weeks. Participants not meeting this NICE criterion returned to routine treatment under the care of their usual Clinical Team. Following assessment at week 48, participants meeting the NICE criteria of adequate response were eligible to continue on study treatment for a further 24 weeks. Participants not meeting this NICE criterion returned to routine treatment under the care of their usual Clinical Team.
Arm/Group | Secukinumab (AIN457) 150mg | Secukinumab (AIN457) 300mg
Serious Adverse Events (participants affected / at risk) | 14/115 | 24/179
Other Adverse Events (participants affected / at risk) | 88/115 | 152/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (AIN457) 150mg (N=115) | Secukinumab (AIN457) 300mg (N=179)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chills (General disorders) | 0 | 1
Electrocution (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2
H1N1 influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Alcoholic seizure (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Drug withdrawal convulsions (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 0 | 1
Glomerulonephritis proliferative (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Pregnancy of partner (Social circumstances) | 0 | 1
Diabetic macroangiopathy (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (AIN457) 150mg (N=115) | Secukinumab (AIN457) 300mg (N=179)
Dry eye (Eye disorders) | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 14 | 16
Dyspepsia (Gastrointestinal disorders) | 7 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4
Mouth ulceration (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 2 | 19
Toothache (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 6 | 12
Chest discomfort (General disorders) | 3 | 0
Fatigue (General disorders) | 9 | 8
Influenza like illness (General disorders) | 8 | 7
Seasonal allergy (Immune system disorders) | 3 | 6
Cellulitis (Infections and infestations) | 0 | 4
Conjunctivitis (Infections and infestations) | 2 | 7
Ear infection (Infections and infestations) | 7 | 7
Folliculitis (Infections and infestations) | 1 | 4
Gastroenteritis (Infections and infestations) | 3 | 3
Influenza (Infections and infestations) | 5 | 9
Lower respiratory tract infection (Infections and infestations) | 6 | 14
Nasopharyngitis (Infections and infestations) | 27 | 52
Oral candidiasis (Infections and infestations) | 2 | 7
Oral herpes (Infections and infestations) | 6 | 5
Otitis externa (Infections and infestations) | 3 | 2
Pharyngitis (Infections and infestations) | 1 | 5
Sinusitis (Infections and infestations) | 3 | 12
Tinea pedis (Infections and infestations) | 1 | 4
Tonsillitis (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 8 | 9
Urinary tract infection (Infections and infestations) | 4 | 10
Viral upper respiratory tract infection (Infections and infestations) | 6 | 11
Vulvovaginal candidiasis (Infections and infestations) | 6 | 8
Contusion (Injury, poisoning and procedural complications) | 2 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 7
Joint injury (Injury, poisoning and procedural complications) | 3 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 4
Alanine aminotransferase increased (Investigations) | 2 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 5
Blood creatine phosphokinase increased (Investigations) | 3 | 6
Blood glucose increased (Investigations) | 4 | 3
Blood triglycerides increased (Investigations) | 2 | 4
Gamma-glutamyltransferase increased (Investigations) | 1 | 7
Lipase increased (Investigations) | 1 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0
Gout (Metabolism and nutrition disorders) | 3 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 19
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 16
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 11
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 9
Dizziness (Nervous system disorders) | 2 | 9
Headache (Nervous system disorders) | 27 | 28
Lethargy (Nervous system disorders) | 3 | 5
Migraine (Nervous system disorders) | 4 | 2
Paraesthesia (Nervous system disorders) | 3 | 2
Depression (Psychiatric disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 29
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 3 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4
Intertrigo (Skin and subcutaneous tissue disorders) | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 15 | 28
Rash (Skin and subcutaneous tissue disorders) | 4 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.